CLINICAL TRIAL: NCT03148925
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Pharmacodynamics of Increasing Subcutaneous Doses of SELA-070 in Healthy Adult Smokers
Brief Title: Safety and Pharmacodynamcis of SELA-070 Nicotine Vaccine in Smokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Selecta Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SELA-070/101; 2017-000534-65 (EudraCT Number)
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-09

CONDITIONS: Smoking Cessation
Keywords: nicotine vaccine; smoking vaccine; smoking cessation; SELA-070
MeSH Terms: conditions — Smoking Cessation | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SELA-070 (Experimental)
  Interventions: Biological: SELA-070
- Saline (Placebo Comparator)
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: SELA-070 — Sub-cutaneous injection, multiple dose
  Arms: SELA-070
Biological: Saline — Sub-cutaneous injection, multiple dose
  Arms: Saline

SUMMARY:
The purpose of this study is to evaluate the safety and pharmacodynamics of SELA-070. Increasing subcutaneous doses of SELA-070 will be administered to healthy smoker volunteers. The resulting safety profile and anti-nicotine antibody levels will be evaluated.

ELIGIBILITY:
Primary Inclusion Criteria:

* Healthy Smokers
* Subjects must smoke a minimum of 10 but not more than 25 cigarettes per day for at least 3 months prior to enrollment
* Written informed consent

Primary Exclusion Criteria:

* Prior exposure to nicotine vaccines
* Female subjects of childbearing potential
* Current use of immunosuppressive agents
* History of or current autoimmune disorder of immunosuppressive condition (e.g. HIV infection)
* Concurrent participation or participation within 8 weeks prior to the initial study drug administration in a drug/device or biologic investigational research study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2018-10-18 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of multiple subcutaneous injections of SELA-070 as assessed by frequency of vaccine related adverse events, graded by severity | 21 weeks

SECONDARY OUTCOMES:
Immunogenicity of SELA-070 by measuring anti-nicotine antibody titers by Enzyme-Linked Immunosorbent Assay (ELISA). | 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lucardie, MD, Principal Investigator — SGS LSS Clinical Pharmacology Unit - Antwerpen
Locations (1):
- SGS LSS Clinical Pharmacology Unit, Antwerp, Belgium